CLINICAL TRIAL: NCT01341756
Title: Palliative Radiotherapy for Symptomatic Locally Advanced Gastric Cancer: A Phase II Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Jeremy Tey, National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B/09/134
Record Dates: First submitted 2011-04-18; First posted 2011-04-26 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-04

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Radiotherapy; palliation; bleeding; pain; obstruction
MeSH Terms: conditions — Stomach Neoplasms; Hemorrhage; Pain; Bites and Stings | interventions — Palliative Care; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy for gastric cancer (Experimental): Single arm study
  Interventions: Radiation: Palliative Radiotherapy

INTERVENTIONS:
Radiation: Palliative Radiotherapy — Palliative Radiotherapy to a total dose of 36Gy in 12 fractions
  Other Names: palliation, radiotherapy

SUMMARY:
The hypothesis of this study is that a radiotherapy dose of 36Gy in 12 fractions, which equates to a BED of 48.6Gy, increases the response rates of symptom relief compared to historical controls.

DETAILED DESCRIPTION:
The hypothesis of this study is that a radiotherapy dose of 36Gy in 12 fractions, which equates to a BED of 48.6Gy, increases the response rates of symptom relief compared to historical controls. (Tey et al.) With this dose fractionation is used for bleeding, there is an increase in response rates from 55%(historical) to 75%for pain, there is an increase in response rates from 25% (historical) to 45% for obstruction, there is an increase in response rates from 25% (historical) to 45%

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the stomach
* Treated with palliative intent
* At least one index symptom such as bleeding, obstruction or pain
* No prior abdominal radiotherapy
* Not on chemotherapy

Exclusion Criteria:

* Patients treated with radical intent
* Previous abdominal radiotherapy
* Patients on chemotherapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Response of bleeding to radiotherapy | At the 12th fraction of radiotherapy and at one month post radiotherapy
  Percentage of patients who do not require blood transfusion after radiotherapy

SECONDARY OUTCOMES:
Number of patients who develop anorexia, nausea, vomiting as per common toxicity criteria v3.0 | within the first 14 days from start of radiotherapy
  Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Tey, FRANZCR, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Tey J, Zheng H, Soon YY, Leong CN, Koh WY, Lim K, So JBY, Shabbir A, Tham IWK, Lu J. Palliative radiotherapy in symptomatic locally advanced gastric cancer: A phase II trial. Cancer Med. 2019 Apr;8(4):1447-1458. doi: 10.1002/cam4.2021. Epub 2019 Feb 20. PMID 30790469